CLINICAL TRIAL: NCT02117960
Title: Assessing the Effects of Omega-3 Supplementation on Serum HSP27, HSP70, YKL40, BMP-4 Levels in Male Patient With Coronary Artery Disease
Brief Title: Assessing the Effects of Omega-3 Supplementation on Serum HSP27, HSP70, YKL40, BMP-4 Levels in Male Patient With CAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2486
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Cardiovascular Disease
Keywords: atherosclerotic; BMP-4; YKL40; HSP70; HSP27
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CVD, Omega-3 (Active Comparator): patients with Cardiovascular disease who receive 4g/d omega-3
  Interventions: Dietary Supplement: Omega-3
- CVD, Placebo (Placebo Comparator): patients with cardiovascular disease who receive 4 cap of placebo/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 — 4 cap 1 g Omega-3 per day for 2 months
  Other Names: n-3 fatty acids; n-3 PUFA
  Arms: CVD, Omega-3
Dietary Supplement: Placebo — 4 cap 1 g Placebo(paraffin) per day for 2 months
  Arms: CVD, Placebo

SUMMARY:
The aim of this study is the comparison between the effects of supplementation with omega 3 or placebo for 8 weeks in serum level of BMP-4, YKL40, HSP70, HSP27 in patients with cardiovascular disease.

DETAILED DESCRIPTION:
The aim of this study is the comparison between the effects of supplementation with omega 3 or placebo for 8 weeks in serum level of BMP-4, YKL40, HSP70, HSP27 in patients with cardiovascular disease. In this randomized, double-blind clinical trial, placebo-controlled, single-center, and phase two trials, 42men aged 45-65 years with Coronary Artery Disease are enrolled in the study from Tehran Heart Center. After signing informed consent all individuals complete a general information form , 24-hour food recall for 3 days will be taken from the participants at the beginning and the end of the study,. Selected samples are randomly classified into 2 blocks of groups receiving supplement and placebo. The supplement group, will receive 4 g/day omega 3 fatty acid for 8 weeks and the placebo group will also receive placebo (containing 4 g of edible paraffin) (similar in terms of color, shape and size). Patients are recommended to sustain their diets and medication dose (s) during the study and also advised to maintain a constant level of physical activity. Blood samples will be collected after 8-12 hours fasting and anthropometric variables, biochemical parameters and physical activity before and after the trial will be measured.

ELIGIBILITY:
Inclusion Criteria:

* CVD patients 45- 65 years old, patients with ≥ 50% stenosis in at least one coronary angiogram demonstrated, body mass index in the range 18.5- 35, avoidance of dietary supplements, vitamins and herbal products at least 3 months before and throughout the intervention, willingness to participation,

Exclusion Criteria:

* people who have used omega 3 supplements in last 3 months, having chronic renal disease , GI disease, hepatobiliary diseases, hematological disorders, hypo- or hyperthyroidism, Smokers

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Serum Heat Shock Protein 70(HSP70) | Change frome baseline at 2 months

SECONDARY OUTCOMES:
Serum Ox-LDL | Change frome baseline at 2 months
Serum BMP4 (Bone Morphogenic Protein4) | Change frome baseline at 2 months
Serum Heat Shock Protein 27(HSP27) | Change frome baseline at 2 months
Serum YKL40 | Change frome baseline at 2 months
Serum hsCRP | Change frome baseline at 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Jalali, Ph.D, Study Director — Department of Nutrition & Biochemistry, School of Public Health, Tehran University of Medical Sciences (TUMS)
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran